CLINICAL TRIAL: NCT06700135
Title: Efficacy of Sensorimotor Stimulation on Oral Feeding Skills for Neonates Post Hypoxic Ischemic Encephalopathy in Neonatal Intensive Care Unit
Brief Title: Sensorimotor Stimulation on Oral Feeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed fekry ibrahim salman, assistant professor, Al-Ahliyya Amman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sensorimotor stimuli
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Neonates Post Hypoxic Ischemic Encephalopathy
Keywords: Neonates; Hypoxic ischemic encephalopathy; Sensorimotor stimulation
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): the control group, which comprised 15 neonates, received only traditional medical treatment.
  Interventions: Other: sensorimotor stimulation program sessions
- study group (Experimental): The study group, consisting of 15 neonates, received traditional medical treatment along with sensorimotor stimulation program sessions. These sessions included oral stimulation protocol, Tactile/Kinesthetic (T/K) intervention, feeding position, and oral support.
  Interventions: Other: sensorimotor stimulation program sessions

INTERVENTIONS:
Other: sensorimotor stimulation program sessions — The study group, consisting of 15 neonates, received traditional medical treatment along with sensorimotor stimulation program sessions. These sessions included oral stimulation protocol, Tactile/Kinesthetic (T/K) intervention, feeding position, and oral support.

SUMMARY:
Background: Perinatal asphyxia and the resulting hypoxic-ischemic encephalopathy (HIE) are significant causes of irreversible adverse neurodevelopmental outcomes in children. Neonates and infants with HIE commonly experience difficulties in learning the oromotor skills of sucking, swallowing, and breathing. These feeding problems can lead to severe complications such as weight loss, dehydration, malnutrition, and developmental deficits.

Objective: The study aims to assess the efficacy of sensorimotor stimulation intervention on oral skills in neonates with post-hypoxic ischemic encephalopathy in the neonatal intensive care unit (NICU).

Methods: The study will include thirty infants with hypoxic-ischemic encephalopathy. They will be divided into two equal groups: The study group receive traditional medical treatment as well as a sensorimotor stimulation program, whereas the control group receive only traditional medical treatment

ELIGIBILITY:
Inclusion Criteria:

* neonates, diagnosed with post-hypoxic ischemic encephalopathy

Exclusion Criteria:

* Neonates with congenital anomalies affecting the oral-facial area,
* or syndromes associated with developmental delays,
* chronic medical complications

Ages: 1 Day to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-11-28 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
Transition time from tube to full oral feeding | - At least one-time breast feeding in a 24-hour period (Fucile et al., 2013). - Consuming eight feedings per day for two consecutive days. - Capable of consuming orally over 80% of the recommended total fluid intake within a 24-hour period (Premji et
  the number of days from the commencement of the intervention to the first day of exclusive oral feeding.
Time taken to accomplish exclusive oral feeding | At least one-time breast feeding in a 24-hour period (Fucile et al., 2013). - Consuming eight feedings per day for two consecutive days. - Capable of consuming orally over 80% of the recommended total fluid intake within a 24-hour period (Premji et a
  this is the number of days from the beginning of oral feeding until discharge.

SECONDARY OUTCOMES:
Total hospital stay | At least one-time breast feeding in a 24-hour period (Fucile et al., 2013). - Consuming eight feedings per day for two consecutive days. - Capable of consuming orally over 80% of the recommended total fluid intake within a 24-hour period
  this is the number of days from the start of the oral stimulation program until discharge from the NICU.

IPD SHARING:
Plan to Share IPD: No